CLINICAL TRIAL: NCT00241475
Title: An Open Label, Non-Comparative, Phase II Study of ZD1839 (Iressa) as First-Line Treatment in Subjects With Relapsed Prostate Cancer Following Radical Prostatectomy or Radiotherapy
Brief Title: Gefitinib in the Treatment of the First Relapse of Prostate Cancer Beyond Prostatectomy or Radiotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0155
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Prostate Cancer
Keywords: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
To evaluate activity of gefitinib in subjects with relapsed prostate cancer by estimating PSA response rate at study closure

ELIGIBILITY:
Inclusion Criteria:

* Relapsed prostate cancer after prostatectomy or radiotherapy
* PSA levels below 10 ng/mL
* Lymph node negative
* Metastasis negative
* Withdrawal of hormone therapy at least 6 months before entry into the study
* Written informed consent

Exclusion Criteria:

* Metastatic disease
* Hormonal treatment 6 months before study entry
* Concomitant radiotherapy, surgery and/or chemotherapy
* ILD

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-12; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
PSA response rate at statistical study closure based on the percentage of subjects experiencing PSA normalization or a > 50% reduction in PSA levels compared with study entry sustained for 3 months (i.e. three consecutive measurements)

SECONDARY OUTCOMES:
TTF (failure defined as a need for additional/alternative therapy due to PSA progression, metastases or AEs)
Duration of PSA response
PFS (progression defined as doubling in PSA levels compared with the PSA level at study entry)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Finland Medical Director, MD, Study Director — AstraZeneca Finland
Locations (1):
- Research Site, Helsinki, Finland